CLINICAL TRIAL: NCT06109467
Title: A Phase II Study Of Neratinib In Combination With Chemotherapy/Trastuzumab/Pembrolizumab In HER2 Overexpressing Gastroesophageal Cancers
Brief Title: Neratinib In Combination With Chemotherapy/Trastuzumab/Pembrolizumab In HER2 Gastroesophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Puma Biotechnology, Inc. (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21917
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: GastroEsophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — neratinib; Trastuzumab; Oxaliplatin; Fluorouracil; Leucovorin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with Neratinib with Trastuzumab, Pembrolizumb and mFOLFOX (Experimental): All patients will be treated with combination of neratinib with trastuzumab, pembrolizumab and mFOLFOX. All patients will receive standard dose 5FU/oxaliplatin/trastuzumab every 2 weeks. Pembrolizumab 400 mg intravenously will be administered once every 6 weeks. Neratinib will be dosed 240 mg orally daily
  Interventions: Drug: Neratinib; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: 5-Fluorouracil + leucovorin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Neratinib — All participants will take 240mg neratinib by mouth every day beginning cycle 1 day 1.
  Other Names: NERLYNX
Drug: Trastuzumab — All participants will receive standard dosing (6mg/kg loading dose, 4 mg/kg subsequent doses) of Trastuzumab by IV infusion day 1 of each 2 week cycle.
  Other Names: Herceptin
Drug: Oxaliplatin — All participants will receive 85mg Oxaliplatin by IV infusion day 1 of each 2 week cycle.
  Other Names: Eloxatin
Drug: 5-Fluorouracil + leucovorin — All participants will receive 400 mg/m^2 5-Fluorouracil (5FU)+ 400 mg/m^2 leucovorin day 1 of each 2 week cycle; 5FU continuous infusions on days 1 and 2 of each 2 week cycle. (5FU + leucovorin may be eliminated from regimen per PI discretion)
Drug: Pembrolizumab — All participants will receive 400mg Pembrolizumab by IV infusion day 1 of every 3rd 2 week cycle.
  Other Names: Keytruda

SUMMARY:
The purpose of the study is to test the effects, both good and bad, of the research study drug Neratinib in combination with Trastuzumab, Pembrolizumab and FOLFOX chemotherapy. This study will also look at the safety of Neratinib in combination with Trastuzumab, Pembrolizumab and FOLFOX in HER2 overexpressing Gastroesophageal cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically confirmed esophageal, gastric or gastroesophageal junction (GEJ) adenocarcinoma by the enrolling institution.
* Patients must have esophageal, gastric or GEJ adenocarcinoma with HER2 overexpression and/oramplification as determined by immunohistochemistry (IHC 3+) or fluorescent in situ hybridization (FISH+ as defined as HER2:CEP17 ratio ≥2.0 if IHC 2+). No central testing will be required. The testing can be performed on archival tissue that is less than 6 months old. If archival tissue is more than 6 months old, a new biopsy must be obtained to confirm HER2 status prior to enrollment.
* Patients may have received no prior chemotherapy or be treatment naïve for stage IV disease. Patients may have received prior adjuvant therapy (chemotherapy and/or chemoradiation) if more than 6 months have elapsed between the end of adjuvant therapy and expected date of treatmentstart on this study. Patients who have received maintenance nivolumab after chemoradiation and surgery would be eligible as long as the last dose of nivolumab was more than 3 months from thedate of expected date of treatment start on this study.
* Patients must have measurable disease per RECIST v1.1.
* Patients must not have active decompensated cardiomyopathy and must have a normal LVEF (≥ 53%). If a patient has a borderline LVEF (40-52%), they may be considered after consultation with cardiology and study PI.
* ECOG performance status 0 or 1.
* Demonstrate adequate organ function as outlined in protocol.
* Female patients of childbearing potential should have a negative urine or serum pregnancy within 72hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 2 years.
* Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system- (CNS-) directed therapy shows no evidence of progression at 4-6 weeks after treatment.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational treatment within 4 weeks of the first dose of treatment.
* Has had prior chemotherapy, targeted small molecule therapy, immunotherapy prior to study Day 1 for metastatic disease or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent with the exception of alopecia or immune mediated hypothyroidism.

Note: (a) If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. (b.) If patient received radiation treatment for brain metastases, then it should have completed more than 6 weeks prior to starting Day 1 of treatment.

* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic therapy in the past 2 years (i.e. disease modifying agents, immunosuppressants or corticosteroids). Replacement therapy (i.e. thyroxine, insulin, physiologic doses of corticosteroids for adrenal or pituitary insufficiency etc.) is not considered a form of systemic therapy and is allowed.
* Has a diagnosis of immunodeficiency or receives chronic steroid therapy (in doses exceeding prednisone 10 mg/day equivalent).
* Has history of non-infectious pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has baseline neuropathy > grade 1.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has had COVID-19 infection within 90 days of confirming eligibility or has sequelae of COVID-19 infection such as symptoms that cannot be explained by any other medical event or comorbidity.
* Vaccination for COVID-19 is allowed on the study unless patient had a grade 3 event after either dose of the vaccine and has not resolved to grade 1 before registration.
* Is unwilling to give written informed consent, unwillingness to participate, or inability to comply with the protocol for the duration of the study.
* Has active or clinically significant cardiac disease including: (a.) Congestive heart failure - New York Heart Association (NYHA) > Class II. (b) Active coronary artery disease.(c) Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.(d) Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before initiation, or myocardial infarction within 6 months before initiation. (e) QTc interval >450 ms for men or >470 ms for women or known history of QTc prolongationor Torsades de Pointes.
* Patient has significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g.,Crohn's disease, malabsorption, or Grade ≥2 (NCI CTCAE v.5.0) diarrhea of any etiology at screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  ORR is defined as the best overall response as complete response (CR) + partial response (PR) per RECIST v1.1 criteria. As per RECIST 1.1 criteria, any evidence of response in measurable lesions will be counted toward the calculation of ORR.ORR will be calculated through exact binomial distribution with a 2-sided 95% CI among patients who obtain at least one dose of study drug.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Up to 24 months
  CBR is defined as complete response + partial response + stable disease per RECIST v1.1 criteria. CBR will be calculated through exact binomial distribution with a 2-sided 95% CI among patients who obtain at least one dose of study drug.
Duration of Response | Up to 24 months
  Duration of response will be calculated from the time of first response (complete response or partial response) until disease progression or death, whichever comes first. Duration of response will be summarized descriptively using Kaplan Meier medians and quantities.
Overall Survival (OS) | Up to 24 months
  OS will be calculated from start of study treatment to death due to any cause. Overall survival will be summarized descriptively using Kaplan Meier medians and quantities.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Won Kim, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided